CLINICAL TRIAL: NCT00791362
Title: Effects and Costs of a National Continuous Improvement Programme on Cardiovascular Diseases in Primary Care
Brief Title: Evaluation Research of a National Accreditation and Improvement Programme for General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PAHVZ; 170883001
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2012-05

CONDITIONS: Cardiovascular Disease
Keywords: accreditation; cardiovascular disease; primary care
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Accreditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- improvement programme CVD (Other)
  Interventions: Other: National programme for accreditation and improvement of GP
- improvement programme other conditions (Other)
  Interventions: Other: National programme for accreditation and improvement of GP

INTERVENTIONS:
Other: National programme for accreditation and improvement of GP — The national programme for accreditation and improvement of general practice. This procedure consists of a package of activities, including audit, feedback, improvement plans, and follow-up. It is partly based on new theories on quality improvement, including the use of market forces and pressure for accountability. For the purpose of the study, the intervention group will be requested to focus their improvement plans in the first year on cardiovascular diseases. The control group is requested to focus their improvement plans in the first year on other domains and to provide cardiovascular care as usual.

SUMMARY:
Objective: This study aims to determine the effectiveness and efficiency of a national accreditation and improvement programme for general practice, focusing on patients with established cardiovascular diseases.

Design: Cluster randomised trial with a block design. All practices start with the accreditation procedure.Intervention group practices are requested to focus their improvement plans in the first year on cardiovascular disease. Control group practices are requested to focus their improvement plans in the first year on other domains. Measurements at baseline are based on the standard audit in the accreditation procedure. Follow-up measurements are done 12 months after approval of improvement plans.

Participants: Primary care physicians in The Netherlands.

Interventions to be implemented: improvement plans concerning cardiovascular risk management, as described by recently updated national multidisciplinary evidence-based NHG / CBO guidelines, considering patients with established cardiovascular diseases.

Implementation strategy: The national programme for accreditation and improvement of general practice. This procedure consists of a package of activities, including audit, feedback, improvement plans, and follow-up.

Outcome measures: Primary outcomes are percentages of patients with CVD who have acceptable systolic blood pressure and cholesterol levels (quantified according to the indicators in the accreditation)and who use aspirin or alternatives. Secondary measures include clinical and organisational indicators of quality of cardiovascular care, such as percentages of patients with cardiovascular disease whose risk factors were assessed and who received specific medication.

Economic evaluation: Incremental cost effectiveness ratio's are determined of the implementation strategy compared to no implementation. The analysis will take a societal perspective and a time horizon of the observed period as well as a hypothetical 10 years period (using modelling). Uncertainty related to the estimations is examined with sensitivity analyses and bootstrapping. The long term economic evaluation is based on Markov modelling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established cardiovascular diseases (myocard infarct, angina pectoris, cerebrovascular accident, Transient Ischaemic Attack, peripheral vascular disease, aneurysma aortae)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1685 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentages of patients with CVD who have acceptable systolic blood pressure and cholesterol levels (quantified according to the indicators in the accreditation)and who use aspirin or alternatives. | dec 2008-feb 2011

SECONDARY OUTCOMES:
Clinical and organisational indicators of quality of cardiovascular care, such as percentages of patients with cardiovascular disease whose riskfactors were assessed and who received specific medication. | dec 2008-feb 2011

CONTACTS AND LOCATIONS:
Overall Officials: Michel Wensing, Dr, Principal Investigator — IQ Scientific Institute for Quality of HealthCare - UMC St Radboud
Locations (1):
- 23 Locations, Nijmegen, Netherlands

REFERENCES:
- [Derived] Nouwens E, van Lieshout J, Bouma M, Braspenning J, Wensing M. Effectiveness of improvement plans in primary care practice accreditation: a clustered randomized trial. PLoS One. 2014 Dec 2;9(12):e114045. doi: 10.1371/journal.pone.0114045. eCollection 2014. PMID 25463149
- [Derived] Nouwens E, Van Lieshout J, Adang E, Bouma M, Braspenning J, Wensing M. Effectiveness and efficiency of a practice accreditation program on cardiovascular risk management in primary care: study protocol of a clustered randomized trial. Implement Sci. 2012 Oct 4;7:94. doi: 10.1186/1748-5908-7-94. PMID 23035760